CLINICAL TRIAL: NCT05546944
Title: Silicosis-harnessing New Ideas to Conquer the Re-emergence of an Ancient Lung Disease
Brief Title: The SHIELD Study-silicosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Queensland (Other)
Collaborators: The Prince Charles Hospital (Other Government); Royal Prince Alfred Hospital, Sydney, Australia (Other); The Alfred (Other); Austin Hospital, Melbourne Australia (Other)
Responsible Party: Sponsor
Other Study IDs: SHIELD
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-03

CONDITIONS: Silicosis
Keywords: Silicosis; Pneumoconiosis; lung diseases
MeSH Terms: conditions — Silicosis; Pneumoconiosis; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Biomarkers (blood ACE and ferritin)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational cohort study to derive biomarkers which are able to more accurately diagnose silicosis, as well as predict disease progression, assess response to treatment, and hasten therapeutic discovery.

DETAILED DESCRIPTION:
Background: Silicosis is a fatal lung disease caused by inhaling silica particles. Australia is currently facing an epidemic with hundreds of young workers having contracted silicosis from machining engineered stone. AIMS: To establish the SHIELD COHORT and associated SHIELD BIOBANK to drive further discovery including assessing the efficacy of whole lung lavage for accelerated silicosis, uncovering disease biomarkers, and druggable targets.

PARTICIPANTS: 75 participants who are respirable crystalline silica exposed workers, (this includes n=30 with silicosis, n=15 with progressive massive fibrosis and n=30 with no pneumoconiosis). METHODS: Advanced microscopy, 'omic platforms and single cell RNA sequencing. OUTCOME: The SHIELD study builds on the knowledge gap to accurately diagnose silicosis, as well as predict disease progression, assess response to treatment, and hasten therapeutic discovery

ELIGIBILITY:
Inclusion Criteria:

* All workers with a history of significant engineered stone exposure will be potentially eligible.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Respirable crystalline silica (RCS) exposed workers with silicosis or silica induced bronchitis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
the SHIELD study primary outcome is to build up knowledge gap to accurately diagnose silicosis, as well as predict disease progress, assess response to treatment, hasten therapeutic discovery in 12 months. | 12 months
  1. Establish the SHIELD cohort and associated lung fluid, tissue and blood biobank from well phenotyped RCS-exposed workers identified via the screening programs.
  2. Utilise advanced microscopy, 'omic platforms and single cell RNA sequencing (scRNAseq) alongside conventional laboratory techniques, to identify and validate candidate lung and blood biomarkers associated with disease and disease progression at 12 months.
  3. To evaluate associations between baseline characteristics, biomarkers and progression of disease in the full cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Chambers, Principal Investigator — The Prince Charles Hospital
Locations (1):
- The Prince Charles Hospital, Brisbane, Queensland, Australia